CLINICAL TRIAL: NCT06867263
Title: Long-term Evaluation of Patients with Fulguration of Posterior Urethral Valve: a Retrospective Cohort Study
Brief Title: Outcomes of Posterior Urethral Valve Fulguration
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, keroles Ashraf Soliman, Principal Investigator, Assiut University
Other Study IDs: Posterior urthral valve
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Posterior Urethral Valve
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Fulguration — Posterior urethral valve fulguration

SUMMARY:
To evaluate the long-term outcome after fulguration of the posterior urethral valve.

DETAILED DESCRIPTION:
Posterior Urethral Valves (PUV) are the most common cause of lower urinary tract obstruction. More severe forms are detected early in pregnancy (mainly type I), while other forms are usually discovered later in childhood when investigating lower urinary tract symptoms. Bladder dysfunction is common and is associated with urinary incontinence in about 55% (0%-72%). Despite the removal of the obstruction by urethral valve ablation, pathological changes in the urinary tract can occur with progressive bladder dysfunction, which can cause deterioration of the upper urinary tract as well. For this reason, all children with PUV require long-term follow-up, always until puberty. In many cases, the life-long current status is uncertain. The current literature lacks research on long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fulguration of PUV since 1 year or more

Exclusion Criteria:

* Patients with neurogenic bladder or meningocele or spina bifida .

Patients with renal parenchymal disease and inflammation not related to posterior urethral valve .

Diabetic patients .

Parental refusal .

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and children
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The rate of spontaneous voiding with insignificant or absent PMR ( according to equation to age ) after one year from fulguration of the PUV. | One year postoperative

REFERENCES:
- [Background] Hennus PM, de Kort LM, Bosch JL, de Jong TP, van der Heijden GJ. A systematic review on the accuracy of diagnostic procedures for infravesical obstruction in boys. PLoS One. 2014 Feb 20;9(2):e85474. doi: 10.1371/journal.pone.0085474. eCollection 2014. PMID 24586242
- [Background] Malin G, Tonks AM, Morris RK, Gardosi J, Kilby MD. Congenital lower urinary tract obstruction: a population-based epidemiological study. BJOG. 2012 Nov;119(12):1455-64. doi: 10.1111/j.1471-0528.2012.03476.x. Epub 2012 Aug 24. PMID 22925164